CLINICAL TRIAL: NCT02397746
Title: Post Market Clinical Follow-Up Study Protocol for PROFEMUR® Gladiator Cemented Femoral Stems
Status: Terminated | Type: Observational
Why Stopped: Research site unable to support further study requirements
Sponsor: MicroPort Orthopedics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 12-LJH-002J
Record Dates: First submitted 2015-03-19; First posted 2015-03-25 (Estimated); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Joint Disease
Keywords: osteoarthritis; avascular necrosis; ankylosis; protrusio acetabuli; rheumatoid arthritis; correction of functional deformity; revision procedures
MeSH Terms: conditions — Joint Diseases; Osteoarthritis; Osteonecrosis; Ankylosis; Arthritis, Rheumatoid | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Total Hip Arthroplasty: Single group previously implanted with the following combination of components: PROFEMUR® Gladiator femoral stem, MicroPort acetabular shell, MicroPort Orthopedics polyethylene or ceramic liner, MicroPort Orthopedics metal or ceramic femoral head.
  Interventions: Device: total hip arthroplasty implant

INTERVENTIONS:
Device: total hip arthroplasty implant
  Other Names: PROFEMUR Gladiator femoral stem

SUMMARY:
MicroPort Orthopedics (MPO) is conducting this post market clinical follow-up (PMCF) study to evaluate the safety and efficacy of its total hip arthroplasty (THA) European Union (EU) . These types of studies are required by regulatory authorities for all THA devices that do not have clinical evidence available at the time of gaining approval to market in the EU. This study has been designed in accordance with MEDDEV 2.12/2 rev 2.

DETAILED DESCRIPTION:
Total hip arthroplasty (THA) has been performed since the early 1920s and is generally considered to be one of the most successful orthopaedic surgeries performed. The 8th Annual Report from the National Joint Registry of England and Wales reported 95.3% component survivorship at 7 years for over 300,000 THA implantations. MicroPort Orthopedics, Inc. (MPO) currently markets several THA components throughout the world, including the European Union (EU). As part of the process for gaining approval to market in the EU, MPO is conducting this post market clinical follow-up (PMCF) study to evaluate the safety and efficacy of these THA components. The objectives of this study are to evaluate component survivorship and total functional outcome scores of implanted subjects at out to 10 years follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Has undergone primary THA for any of the following:
* Non-inflammatory degenerative joint disease such as osteoarthritis, avascular necrosis, ankylosis, protrusio acetabuli, or painful hip dysplasia;
* Inflammatory degenerative joint disease such as rheumatoid arthritis; or
* Correction of functional deformity
* Subject is implanted with the specified combination of components
* Subject is willing and able to complete required study visits or assessments

Exclusion Criteria:

* Subjects implanted with a metal-on-metal articulation
* Subjects implanted with non-MPO or non-Wright Medical Technology components (femoral heads, acetabular shells, acetabular liners) in the enrolled THA
* Subjects skeletally immature (less than 21 years of age) at time of primary THA surgery
* Subjects currently enrolled in another clinical study which could affect the endpoints of this protocol
* Subjects unwilling to sign the Informed Consent document
* Subjects with substance abuse issues
* Subjects who are incarcerated or have pending incarceration

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been previously implanted with PROFEMUR® Gladiator femoral stems
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Component Survivorship | 10 years post-operative
  The primary objective of this study is to estimate survivorship of all components at specified intervals out to 10 years follow-up.

SECONDARY OUTCOMES:
Patient functional outcomes | Screening (First Available), 2-5 years, 5-7 years, and 10 years
  To characterize total functional scores, as assessed by Oxford Hip Scores and EQ-5D-3L scores